CLINICAL TRIAL: NCT06354881
Title: Understanding the Relationship Between Controlling Risk Factors and Cerebral Haemodynamic Changes in Lacunar Stroke, and Its Interaction With Ageing
Brief Title: The Relationship Between Controlling Risk Factors and Cerebral Haemodynamics in Lacunar Stroke
Acronym: LACUNAR_CA
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: British Heart Foundation (Other); University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0967; TM61008S3 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2024-03-19; First posted 2024-04-09 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Lacunar Stroke
Keywords: Lacunar; Stroke; Cerebral Autoregulation; Cerebral Blood Flow
MeSH Terms: conditions — Stroke, Lacunar; Stroke | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lacunar Stroke Syndrome Patients: Patients who have been diagnosed with lacunar stroke syndrome. This is a non-intervention study so no intervention will be given. However, the investigators will observe the changes in cerebral haemodynamics of this group before and after they have been given medications to help control hypertension and/or diabetes which are common risk factors of lacunar stroke syndrome.
  Interventions: Device: Transcranial Doppler Ultrasonography (TCD) during sit-stand manoeuvres

INTERVENTIONS:
Device: Transcranial Doppler Ultrasonography (TCD) during sit-stand manoeuvres — TCD will be used to measure the cerebral blood flow in the middle and posterior cerebral arteries. This will be done at rest and during two sit-stand manoeuvres, whereby the participant will be asked to stand (from a seated position) and stay standing for 1 minute. The participant will then be given time to recover before repeating the manoeuvre. This will occur at the first visit and the follow-up visit 4 weeks after.

SUMMARY:
The goal of this observational study is to look at differences in brain blood flow before and after management of risk factors such as high blood pressure and diabetes in patients with lacunar stroke. Participants will be asked to undergo a simple brain blood flow assessment at their initial appointment, whereby they will be asked to sit and stand twice. The patients will then be asked for a follow-up assessment 4 weeks after, identical to the first. This will allow us to look at any changes in brain blood flow from before management of risk factors and 4 weeks after management of risk factors.

DETAILED DESCRIPTION:
Stroke is the second major cause of death across the world leading to high mortality rates and leaving those who experience stroke with a poor quality of life. Lacunar stroke accounts for a quarter of ischemic stroke events and can occur at any age, but is more frequent in the older generation (>65 years) yet not uncommon in younger patients. Lacunar stroke is caused by small vessel disease, whereby occlusions or thrombi occur in the small vessels found deep in the brain structures, around the circle of Willis. This event leads to a decrease in blood supply to certain areas of the brain and damage to surrounding tissues, leaving the brain in a vulnerable state. Further events are then likely to occur such as recurrent stroke, intracranial haemorrhage, additional ischemic events, prolonging symptoms and increasing the risk of damage to the brain. Even though lacunar infarcts occur only in the small vessels of the brain, cognitive impairment is commonly seen post-lacunar stroke emphasising the importance of understanding the trajectory of cerebral haemodynamics after a lacunar infarction. Common treatments involve the use of anticoagulants, antiplatelet therapies (both to stop further blood clots forming), blood pressure (BP) lowering agents (reducing BP to reduce fluctuations in cerebral blood flow) and the management of hyperglycaemia (to help reduce damage to blood vessels).

Cerebral autoregulation (CA) plays a large part in regulating cerebral blood flow (CBF), through maintaining cerebral perfusion, even with fluctuating BP. It does this by regulating the cerebral vasculature through adjustments in vessel diameter. CA has been assessed at rest and challenged with paradigms in healthy volunteers and lacunar stroke patients, however comparisons between younger and older lacunar events incorporating risk factors has not been looked at. The difference in CA phenotype between those with uncontrolled high-risk cardiometabolic factors (often younger patients) and those with moderate/severe small vessel disease and recurrent lacunar stroke syndromes (often older patients) is unknown. Therefore, exploring different risk factors and the different lacunar disease phenotypes is important to identify any differences in cerebral haemodynamics.

Assessing dynamic CA (dCA) in response to fluctuations in BP represents how CA responds to BP fluctuations in the body, allowing better application to the human vasculature, compared to assessing static CA. Multiple paradigms and manoeuvres have been used to assess dCA by inducing a rapid change in BP, but both patient tolerability and ability to measure dCA accurately need to be considered for this study. The sit-stand manoeuvre is a clinically applicable manoeuvre which can be done both in the ward and laboratory with minimal stress to the patient. This manoeuvre has been evaluated in a published review and compared to a thigh-cuff technique which has been used extensively in previous research. The thigh-cuff technique induces a rapid change in arterial blood pressure (ABP) through the rapid deflation of the thigh cuff. However, this repeated action can be painful for some participants making it difficult to apply clinically to frail patients leading to issues of unsuccessful repeats. The review found that autoregulatory index (ARI) values were similar across both the sit-stand and thigh-cuff manoeuvres, showing sit-stand is an accurate manoeuvre to measure CA. The sit-stand manoeuvre was also better tolerated compared to the thigh-cuff.

Following up patients post-stroke as high-risk factors are controlled will help understand changes in CA and could help guide the timing of interventions to manipulate BP and potentially for the impact of rehabilitation programmes.

Lacunar stroke is one of the most common types of stroke, occurring in both younger and older generations. Some studies have observed impaired brain blood flow regulation (cerebral autoregulation) in a cohort of ~57 years of age (median), which has also been seen in those with small vessel disease. Small vessel disease is often seen in older patients who often present with recurrent lacunar strokes despite earlier management of risk factors.

By targeting a younger cohort with uncontrolled risk factors (hypertension and diabetes), the investigators aim to perform a more comprehensive study to investigate the haemodynamic consequences of lacunar strokes in this group. This would be done by using Transcranial Doppler ultrasound (TDC) to measure CBv in patients who are diagnosed with a lacunar stroke and have undiagnosed diabetes and/or hypertension at their initial appointment. To measure a dCA response, the sit-stand manoeuvre will be used. These patients would then receive management of their risk-factors and would be asked to undergo another TCD assessment 4 weeks after their initial appointment. Data would be collected and analysed to look at any differences in cerebral haemodynamics between before and after management of such risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18-120 years.
* Diagnosis of lacunar stroke syndrome.
* New diagnosis or known diagnosis of hypertension and/or diabetes.

Exclusion Criteria:

* Those who lack capacity can have a personal consultee consent to the study if they can still perform study requirements such as the sit-stand manoeuvre. Those who either cannot perform the manoeuvre or do not have a personal consultee to allow them to consent, are not able to take part.
* Those with poorly controlled medical comorbidities affecting cerebral haemodynamics. (eg., heart failure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited from Leicester Royal Infirmary TIA clinic or stroke ward.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood velocity measurements before and after management of uncontrolled risk-factors in those diagnosed with lacunar stroke syndromes. | From enrolment to the end of the follow-up measurements at 4 weeks.
  Absolute values (cm/s) and percentage change (%) in cerebral blood velocity measurements before and after management of uncontrolled risk-factors in lacunar stroke patients.
Arterial blood pressure measurements before and after management of uncontrolled risk-factors in those diagnosed with lacunar stroke syndromes. | From enrolment to the end of the follow-up measurements at 4 weeks.
  Absolute values (mmHg) and percentage change (%) in arterial blood pressure measurements before and after management of uncontrolled risk-factors in lacunar stroke patients.
Heart rate measurements before and after management of uncontrolled risk-factors in those diagnosed with lacunar stroke syndromes. | From enrolment to the end of the follow-up measurements at 4 weeks.
  Absolute values (bpm) and percentage change (%) in heart rate measurements before and after management of uncontrolled risk-factors in lacunar stroke patients.
End-tidal carbon dioxide measurements before and after management of uncontrolled risk-factors in those diagnosed with lacunar stroke syndromes. | From enrolment to the end of the follow-up measurements at 4 weeks.
  Absolute values (mmHg) and percentage change (%) in heart rate measurements before and after management of uncontrolled risk-factors in lacunar stroke patients.
Compare cerebral haemodynamics in lacunar stroke patients with older patients experiencing advanced chronic cerebrovascular disease with lacunar stroke syndromes, whose risk-factors are already managed.(CA). | Data collected from enrolment to the end of the follow-up measurements at 4 weeks. Comparisons to other data and other studies to be done at analysis stage.
  Efficiency of regulatory mechanisms will be analysed through measuring cerebral autoregulation.
Compare cerebral haemodynamics in lacunar stroke patients with older patients experiencing advanced chronic cerebrovascular disease with lacunar stroke syndromes, whose risk-factors are already managed. (VMR). | Data collected from enrolment to the end of the follow-up measurements at 4 weeks. Comparisons to other data and other studies to be done at analysis stage.
  Efficiency of regulatory mechanisms will be analysed through measuring vasomotor reactivity.
Compare cerebral haemodynamics in lacunar stroke patients with older patients experiencing advanced chronic cerebrovascular disease with lacunar stroke syndromes, whose risk-factors are already managed.(ARI). | Data collected from enrolment to the end of the follow-up measurements at 4 weeks. Comparisons to other data and other studies to be done at analysis stage.
  Efficiency of regulatory mechanisms will be analysed through measuring the autoregulatory index.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared, however once analysed and combined (statistically through mean averages etc), the results will be compiled into a report and submitted to a relevant journal, allowing researchers to view them.